CLINICAL TRIAL: NCT01142882
Title: Comparative Effectiveness of Web-based vs. Traditional Adolescent HIV Prevention
Brief Title: Comparative Effectiveness of Web-based Versus Traditional Adolescent HIV Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Lisa A. Marsch, Ph.D., National Development and Research Institutes, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIVPrev613; 1RC1DA028415 (NIH)
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: HIV Infections; Hepatitis; Sexually Transmitted Infections
Keywords: adolescent HIV prevention; web-based interventions; adolescent substance abuse treatment; comparative effectiveness research; HIV prevention; hepatitis prevention; STI prevention
MeSH Terms: conditions — HIV Infections; Hepatitis; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Prevention (Active Comparator): educator-delivered, small-group HIV & disease prevention education
  Interventions: Behavioral: Traditional Prevention
- Web-based Prevention (Experimental): self-directed, interactive & customized web-based HIV & disease prevention education
  Interventions: Behavioral: Web-based Prevention

INTERVENTIONS:
Behavioral: Traditional Prevention — Participants in the traditional prevention intervention condition will complete two sessions (of approx. one hour in duration) across the course of a week, conducted by a trained HIV (and infectious disease) prevention educator; these sessions will typically be conducted in small groups of 2-4 participants but may be offered individually.
  Arms: Traditional Prevention
Behavioral: Web-based Prevention — Participants in the web-based intervention condition will complete an interactive, web-based HIV, hepatitis and STI prevention program. Youth will be asked to complete a customized plan of approximately 2-4 hours in length using the web-based tool; participants will complete two 60-minute sessions per week until they complete their customized plan. Participants can choose to access this intervention using dedicated computer stations set up at their substance abuse treatment setting or can complete these sessions at their own home via the web.
  Arms: Web-based Prevention

SUMMARY:
This study will evaluate the comparative effectiveness and cost-effectiveness of a customized, interactive web-based HIV, sexually transmitted infections (STI) and hepatitis prevention intervention as compared to a traditional, educator-delivered prevention intervention. Both interventions will be offered to youth enrolled in outpatient, community-based substance abuse treatment at our collaborating treatment facilities. Outcomes to be measured include accurate HIV/disease prevention knowledge, intentions to engage in safer sex, actual HIV risk behavior, attitudes toward safer sex and self-reported substance use. The web-delivered intervention under evaluation has the potential to deliver evidence-based content at low cost without increasing demands on treatment staff time or training needs.

DETAILED DESCRIPTION:
This trial will examine the comparative effectiveness and cost-effectiveness of a web-based HIV, hepatitis and STI prevention intervention when offered to youth in outpatient, community-based substance abuse treatment as directly compared to a traditional HIV (and infectious disease) prevention intervention. We will assess the comparative effectiveness and cost-effectiveness of these interventions by primarily examining changes from pre- to post-intervention in accurate HIV/disease prevention knowledge, intentions to engage in safer sex and HIV risk behavior. Additionally, we will examine the extent to which the interventions impact relevant skills acquisition (e.g., communication skills, negotiation skills and condom use skills), attitudes toward safer sex and self-reported substance use, as well as the acceptability of each intervention. We also plan to evaluate youth at both 1 and 3 month post-intervention to examine the durability of effects (including any differential durability of effects across intervention conditions). The web-delivered prevention intervention to be evaluated in this study has the potential to allow for a complex intervention to be delivered at a low cost, without increasing demands on staff time or training needs, and may thereby expand the reach of evidence-based prevention for youth in substance-abuse treatment.

This study will be conducted at three collaborating, community-based adolescent substance abuse treatment programs all of which are housed within the Daytop Village network of services and are located in New York City: (1) Daytop Village's Brooklyn Outreach Center; (2) Daytop Village's Bronx Outreach Center; and (3) Daytop Village's Queens Outreach Center. We expect to recruit approximately one third of the total number of participants from each site.

A total of up to 160 (no fewer than 120) adolescent participants will be enrolled in this study. Participants will be randomly assigned to one of the two study conditions in an intent-to-treat design (n=60-80 per group): (1) computer-delivered intervention or (2) traditional (person-delivered intervention). Participants in the traditional prevention intervention condition will complete two sessions (of approx. one hour in duration) across the course of a week, conducted by a trained HIV (and infectious disease) prevention educator; these sessions will typically be conducted in small groups of 2-4 participants but may be offered individually. Participants in the computer-delivered intervention condition will complete an interactive, web-based HIV, hepatitis and STI prevention program instead of the traditional, person-delivered prevention intervention. Youth will be asked to complete a customized plan of approximately 2-4 hours in length using the web-based tool; participants will complete two 60-minute sessions per week until they complete their customized plan. Participants will access this intervention using dedicated computer stations set up at their substance abuse treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in collaborating adolescent substance abuse treatment program (i.e., Daytop's Brooklyn Outreach Center, Bronx Outreach Center or Queens Outreach Center)
* 12-18 years of age
* Within first 30 days of substance abuse treatment (current treatment episode)
* Not yet received formal HIV prevention intervention during current treatment episode

Exclusion Criteria:

* Plans to move out of the area within the next 5 months
* Insufficient ability to understand and provide informed consent/assent to participate
* Insufficient ability to use English to participate in the consent process, the interventions and/or assessments

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
HIV/disease prevention knowledge | 3 months
behavioral intentions | 3 months
  intentions to engage in safer sex
HIV risk behavior | 3 months
  sexual risk behavior

SECONDARY OUTCOMES:
skills acquisition | 3 months
  communication skills; negotiaion skills & condom use skills
self-reported substance use | 3 months
  as measured via Timeline Follow-back
intervention acceptability | post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Marsch, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.; Honoria M. Guarino, Ph.D., Study Director — National Development and Research Institutes, Inc.
Locations (3):
- United States (3):
  - Daytop Village, Brooklyn Outreach Center, Brooklyn, New York
  - Daytop Village, Queens Outreach Center, Jamaica, New York
  - Daytop Village, Bronx Outreach Center, The Bronx, New York

REFERENCES:
- [Derived] Marsch LA, Guarino H, Grabinski MJ, Syckes C, Dillingham ET, Xie H, Crosier BS. Comparative Effectiveness of Web-Based vs. Educator-Delivered HIV Prevention for Adolescent Substance Users: A Randomized, Controlled Trial. J Subst Abuse Treat. 2015 Dec;59:30-7. doi: 10.1016/j.jsat.2015.07.003. Epub 2015 Jul 15. PMID 26293644